The effect of caudal anesthesia block on perioperative pain control and reduction of the anesthetic agent in pediatric infra-umbilical surgery: A prospective randomized trial

Statistical analysis date 04/04/2022 IRB approval number: 123311219,

## **Study population**

The Consolidated Standards of Reporting Trials (CONSORT) checklist was used for the enrolment and allocation of patients. Children aged between two months and six years who were undergoing infra-umbilical surgeries with ASA PS I were randomly allocated to either group A (GA with CEB) or to group B (GA without CEB)., Both groups were compared based on hemodynamic stability, level of sedation, analgesia need, pain score, and parental satisfaction. Postoperative pain was evaluated by the Children's Hospital Eastern Ontario Pain Scale (CHEOPS), Faces Pain Scale-Revised (FPS-R), and Face, Legs, Activity, Cry CONSOL ability (FLACC) scales The raw data which was collected from case report forms were entered into a Microsoft Excel Spreadsheet initially. Then, the data have been transferred to and analyzed by IBM SPSS Statistics software version 21. The categorical and numerical variables of both groups were analyzed and compared. Data are expressed as n (%), mean  $\pm$  standard deviation or median and interquartile range (IQR) according to distribution normality. Continuous variables were compared using the Mann-Whitney U test, and categorical variables were compared using Fisher's exact test or Pearson Chi-square test. P < 0.05 was considered statistically significant. The confidence interval was set at 95%.

## **Tables and Figure legends**

**Table 1.** Demographic parameters of children with (group A) or without (group B) caudal block anesthesia.

| Demographic parameters | Group A (n=36) | Group B (n=36) | P |
|-----------------------------|----------------|-----------------|-----|
| Age (months), mean $\pm$ SD | 20.68 ±1.7 | 29,688 ± 3.4 | 0.3 |
| Sex Female | 16 (13%) | 15 (11.25%) | 0.5 |
| Male | 20 (15%) | 21(15.75%) | |
| Heights (cm), mean $\pm$ SD | $90\pm2.08$ | $103 \pm 4{,}2$ | 0.8 |
| Weights (kg), mean $\pm$ SD | 9 ± 1,05 | $12\pm3,\!02$ | 0.6 |

SD= standard deviation.

**Table 2.** Differences between children with or without caudal block anesthesia in the average pain scores at the various time points according to Children's Hospital Eastern Ontario Pain Scale (CHEOPS).

| Variables | Group A (n=36) | Group B (n=36) | P |
|----------------------|-----------------|-----------------|----------|
| CHEOPS Score average | $3 \pm 0.11$ | 5 ± 0.49 | < 0.005 |
| At 30 minutes | $2.6 \pm 0.41$ | $4\pm0.44$ | < 0.003 |
| At 1 hour | $2.11\pm0.98$ | $4\pm0.54$ | < 0.0001 |
| At 2 hours | $3 \pm 0.44$ | $4\pm0.65$ | < 0.003 |
| At 6 hours | $3.05 \pm 1.53$ | $4.80 \pm 2.04$ | 0.005 |

| Postoperative analgesia | Yes | 3.0 (8.3%) | 36 (100%) | <0.001 |
|-------------------------|---------|------------|------------|---------|
| | No | 33 (91.7%) | 0.0 (0.0%) | |
| Parental satisfaction | Good | 30 (80%) | 5.0 (20%) | < 0.002 |
| | Perfect | 30 (80%) | 5.0 (20%) | < 0.001 |



**Figure 1**. Effect of caudal block versus non-caudal block anesthesia on pain intensity at 1 and 6 hours and the degree of sedation in children undergoing infra-umbilical surgery under general anesthesia.



**Figure 2**. Effect of caudal block versus non-caudal block anesthesia on movement score at 1 and 6 hours postoperatively in children undergoing infra-umbilical surgery under general anesthesia.